CLINICAL TRIAL: NCT05924230
Title: Dose Responsive Study of Ringer's Lactate Solution in Prevention of Post-induction Hypotension Predicted by Inferior Vena Cava Collapsibility Index in Patients Receiving General Anesthesia
Brief Title: Dose Responsive Study of Ringer's Lactate Solution in Prevention of Post-induction Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Abhishek Chatterjee, Consultant, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMH/IEC/JUNE/011/2022
Record Dates: First submitted 2023-04-11; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Post Induction Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RL 10 (Active Comparator): Patients of this group will receive Ringer's lactate (RL) 10ml/kg
  Interventions: Other: RL 10ml/kg
- RL 15 (Active Comparator): Patients of this group will receive 15ml/kg of Ringer's lactate solution
  Interventions: Other: RL 15ml/kg

INTERVENTIONS:
Other: RL 10ml/kg — Inferior vena cava collapsibility index of all patients will be calculated by ultrasonography and if it is >50%, then patients of this group (Group 1) will receive Ringer's lactate 10ml/kg before induction in the receiving area
  Arms: RL 10
Other: RL 15ml/kg — Inferior vena cava collapsibility index of all patients will be calculated by ultrasonography and if it is >50%, then patients of this group (Group 2) will receive Ringer's lactate 15ml/kg before induction in the receiving area
  Arms: RL 15

SUMMARY:
To assess the dose responsiveness of ringer lactate solution in prevention of post-induction hypotension predicted by Ultrasound guided Inferior Vena Cava diameter in patients receiving General anesthesia.

OBJECTIVES Primary - To find the optimum preloading dosage of Ringer Lactate to prevent post induction hypotension.

Secondary - To find the predictive incidence of Post-induction hypotension according to age, gender, type of surgery and comorbidities.

DETAILED DESCRIPTION:
All patients, after Ultrasonographic Inferior vena cava collapsibility index calculation, will receive Lactated Ringer's solution as per body weight and as per their allocated group in the receiving area.

After induction inside the Operating Room, All patients will be monitored continuously using Electrocardiography, pulse oximetry, noninvasive Blood pressure measurement and capnography .

Heart rate, Systolic - Diastolic - Mean blood pressure, Oxygen saturation will be monitored as follows :

1. Baseline parameters - Prior to administration of intravenous Ringer's lactate solution
2. T0 (after administration of intravenous Ringer's lactate solution but prior to induction of anaesthesia),
3. T1-T10 (every minute for first 10 mins after induction of anaesthesia) Our institutional standard practice of induction of Anaesthesia with Fentanyl (2 μg/kg), Propofol (2 mg/kg) and Vecuronium (0.1mg/kg ) will be followed and intubation will be done only after first 10 mins post induction.

Amount of Mephentermine needed to correct hypotension despite RL infusion will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years American Society of Anesthesiologists (ASA) Physical status classification system group I and II Elective surgery under General anesthesia

Exclusion Criteria:

* Age <18 and > 65 American Society of Anesthesiologists (ASA) Physical status classification system group III and IV Systolic blood pressure ≥ 180 mmHg Systolic blood pressure < 90 mmHg Pregnant women Patients with abdominal mass or ascites Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Effective dose of Ringer's lactate solution to prevent post-induction hypotension | 15 months
  This study will try to find out the effective dose of Ringer's lactate solution in ml/Kg that will prevent hypotension after induction of anaesthesia in study population

SECONDARY OUTCOMES:
Effect of age, gender, types of surgery and comorbid conditions on post-induction hypotension | 15 months
  This study will try to find out the effect of age, gender, type of surgery and type of comorbid conditions (like Diabetes, Hypertension etc) on occurence of post-induction hypotension by measuring the % of hypotension in these categories of patients

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Chatterjee, Principal Investigator — Tata Steel
Locations (1):
- Abhishek Chatterjee, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No